CLINICAL TRIAL: NCT04806542
Title: A Mindfulness-based Intervention Improves Resilience, Anxiety, Anger and Disruptive Behaviour in Children With Mental Health Problems: A 2-year Follow-up Study
Brief Title: Two-year Follow-up of a Mindfulness-based Intervention in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TMR-study
Record Dates: First submitted 2021-03-12; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Mental Health Issue
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMR-group (Experimental): 8-week program for schoolchildren called TMR (Training for Resilience and Mindfulness).
  Interventions: Behavioral: TMR-group
- Treatment as Usual (Active Comparator): Individual counselling.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: TMR-group — A mindfulness-based 8 week program.
  Arms: TMR-group
Behavioral: Treatment as usual — Individual counselling.
  Arms: Treatment as Usual

SUMMARY:
The primary aim of this study was to determine whether an 8-week mindfulness-based intervention, called Training for Mindfulness and Resilience (TMR), mitigates moderate mental health symptoms and increases resilience during a 2-year follow-up.

Methods

The participants were 34 schoolchildren in age range of 9-14 years, reporting moderate mental health problems. Participants were randomised into either TMR intervention group (N=22) or control group, receiving best current practice (N=12). The investigators used validated self-rating questionnaires to measure anxiety, depression, anger, disruptive behaviour, self-concept, resilience, stress and mindfulness before treatment with either TMR or control, as well as at 6 months, 1 year and 2 years after treatment period.

ELIGIBILITY:
Inclusion Criteria:

* F32.0 Mild depressive episode
* F32.1 Moderate depressive episode
* F41 Anxiety disorders
* F43 Reactions to stress
* F51 Nonorganic sleep disorders
* F93 Emotional disorders with onset specific to childhood
* F94.8 Other childhood disorders of social functioning
* F94.9 Other childhood disorder of social functioning, unspecified

Exclusion Criteria:

* Ongoing treatment for severe psychiatric disorders (F20-29, F31-F33.3)
* Cognitive disorders
* Difficulties in understanding Swedish
* Neuropsychiatric considerations and diagnosis
* Learning disabilities with difficulties in verbal understanding
* Ongoing parental conflict in conjunction with separation/divorce.
* Attending less than 5 of the 8 sessions of the TMR program.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Anxiety, depression, anger, disruptive behaviour, self-concept according to Beck Youth Inventories. | Change from Baseline anxiety, depression, anger, disruptive behaviour and self-concept at 2 years.
  The investigators used validated self-rating questionnaires called Beck Youth Inventories. Maximum score 300, minimum score 0. Higher values indicate worse outcome except on subscale measuring self-concept where higher score indicate better outcome .
Resilience. | Change from Baseline Resilience at 2 years.
  The investigators used a validated self-rating questionnaire called Resilience Scale 10. Maximum score 40, minimum score 10. Higher values indicate better outcome.
Stress. | Change from Baseline stress at 2 years.
  The investigators used a validated self-rating questionnaire called Stress in Children. Maximum score 92, minimum score 23. Higher values indicate better outcome.
Mindfulness. | Change from Baseline mindfulness at 2 years.
  The investigators used a validated self-rating questionnaire called Child and Adolescent Mindfulness Measure (CAMM). Maximum score 40, minimum score 0. Higher values indicate better outcome.

IPD SHARING:
Plan to Share IPD: No